CLINICAL TRIAL: NCT00624429
Title: A Pilot Study Involving an Asthma Management Program for Inner-city Early Head Start Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Phoenix Children's Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Peggy Radford MD, Phoenix Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-053
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-02

CONDITIONS: Asthma
Keywords: Asthma; Children
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Budesonide respules — Budesonide respules 0.5 mg nebulized once a day for 4 months of the study.
  Other Names: Pulmicort respules

SUMMARY:
The Early Head Start program serves lower socioeconomic inner-city children from birth to 3 years. This population has a higher incidence of asthma due to increased exposures. The primary objective of this study is:

To evaluate the effect of early identification of these high risk, inner-city asthmatic infants, age 1-3 years, and early treatment with pulmicort respules on asthma morbidity (asthma symptoms and use of rescue medications), infant pulmonary functions, and use of health care resources (unscheduled clinic visits, emergency room visits and hospitalizations).

To obtain pilot behavior information using Carey Temperament Scale, Bitsea and expand to Itsea if indicated.

ELIGIBILITY:
Inclusion Criteria:

* Children 12-36 months of age with a history of wheezing or airway reactivity responding to bronchodilators, or diagnosed with asthma by a physician.

Exclusion Criteria:

* Children less than 12 months or greater than 36 months of age.
* Children diagnosed with attention deficit disorder by a physician or psychologist.

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-12 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
FEV0.5 | 2 months and 6 months into study

SECONDARY OUTCOMES:
emergency room visits | number of visits from baseline to 2 months and 2 months to 6months of study
behavior scores | measured at baseline, 2 months and 6 months
number of asthma exacerbations from baseline to 2 months and 2 months to 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Peggy Radford, MD, Principal Investigator — Phoenix Children's Hospital
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States